CLINICAL TRIAL: NCT02071342
Title: Study of ABSORB Stent in Acute Coronary Syndrome
Brief Title: Study of ABSORB Stent in Acute Myocardial Infarction
Acronym: ABSORB-ACS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Umberto I Hospital, Frosinone Italy (Other)
Responsible Party: Principal Investigator, Menichelli Maurizio, Director Division of Cardiology, Umberto I Hospital, Frosinone Italy
Other Study IDs: 350/O/13
Record Dates: First submitted 2014-01-02; First posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Acute Myocardial Infarction; Artery; Deformity, Coronary (Acquired)
Keywords: acute myocardial infarction; bioresorbable vascular scaffold; percutaneous coronary intervention
MeSH Terms: conditions — Congenital Abnormalities | interventions — Angioplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- acute coronary syndrome: patients with acute myocardial infarction who are undergoing coronary angioplasty. MACE at 30 days and 1 year will be assessed . The acute recoil after implantation of bioabsorbable stents will also be assessed
  Interventions: Procedure: angioplasty

INTERVENTIONS:
Procedure: angioplasty — patients with acute coronary syndrome and coronary angioplasty with bioresorbable vascular scaffold.
  Other Names: bioabsorbable everolimus-eluting coronary stent; everolimus-eluting bioresorbable vascular scaffold (BVS)

SUMMARY:
The aim of our study is to evaluate the clinical outcomes at 30 days and 1 year (cardiac death, myocardial infarction, target lesion revascularization (TLR), target vessel revascularization (TVR), thrombosis of the device in patients who are undergoing angioplasty in myocardial infarction and in which bioabsorbable stent was implanted (BVS). Additionally, we will evaluate the acute recoil after implantation of bioabsorbable stents. A 24 months follow-up , by means of coronary angiography accompanied by QCA and assessment with intracoronary ultrasound (IVUS) and VH (virtual histology) is scheduled.

DETAILED DESCRIPTION:
The drug -eluting stents (drug eluting stents , DES) are currently used routinely in the course of coronary angioplasty ( percutaneous coronary intervention , PCI ) and have significantly reduced the incidence of adverse events during follow-up in the medium and long term .

However, the persistence of the metal structure of these devices within the coronary artery over time adds no additional benefit but , on the contrary , it is potentially harmful because it may predispose to coronary thrombosis even after years of implantation, can alter the structure of the vessel for remodeling phenomena, can decrease a coronary vasomotion and reducing the possibilily of a future surgery. The recent development of new devices such as bioabsorbable vascular scaffold " BVS " release of antiproliferative drug ( everolimus ), could provide new clinical advantages especially in patients who are revascularized during acute myocardial infarction. These patients are at higher risk of MACE and stent thrombosis late .

The aim of our study is to evaluate the clinical outcomes conventional to 30 days and 1 year, such as cardiac death, myocardial infarction, target lesion revascularization(TLR ), target vessel revascularization (TVR ), thrombosis of the device in patients who undergo angioplasty in the course of acute coronary syndrome and in which it was implanted bioabsorbable stent ( BVS ). The acute recoil after implantation of bioresorbable vascular scaffold will also be assessed Finally, a follow-up of 24 months we will conduct, by means of coronary angiography accompanied by QCA and IVUS with VH .

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years with acute coronary syndrome (STEMI and NSTEMI) will be enrolled

Exclusion Criteria:

* patients with these characteristics will be excluded: cardiogenic shock (defined as systolic blood pressure less than 80 mmHg for more than 30 minutes or the need for compressors or intravenous-intraaortic balloon counterpulsation), history of bleeding diathesis, history of leukopenia , thrombocytopenia, or severe hepatic or renal dysfunction, a non-cardiac disease associated with a life expectancy of less than one year, participating in another study, or not able to give informed consent due to a prolonged resuscitation cardiopulmonary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute coronary syndrome who are undergoing coronary angioplasty.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
MACE (Death, MI, TLR and TVR) | One year after index procedure
  MACE at 30 days and 1 year (Death, MI, TLR and TVR) and thrombosis of the device in patients with acute coronary syndrome undergoing PCI with stenting bioresorbable

SECONDARY OUTCOMES:
Acute stent Recoil | Within ten minutes after scaffold implantation
  Evaluation of acute recoil after implantation of bioabsorbable stent (BVS).

OTHER OUTCOMES:
conformability | immediately after implantation of the device
  Evaluation of the conformability of the stent and the vessel curvature and angle before and after implantation of the device

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Menichelli, MD, Principal Investigator — Division of Cardiology "Fabrizio Spaziani" Hospital Frosinone, Italy
Locations (1):
- Division of interventional cardiology, Umberto I Hospital, Frosinone, Frosinone, Italy